CLINICAL TRIAL: NCT02969772
Title: Reach and Palmar Grasp in Tetraplegics With Neuromuscular Electrical Stimulation: Assessment and Training.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Enio Walker Azevedo Cacho (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor-Investigator, Enio Walker Azevedo Cacho, PhD, University of Campinas, Brazil
Organization: University of Campinas, Brazil (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06/58891-4
Record Dates: First submitted 2016-11-14; First posted 2016-11-21 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Tetraplegia; Tetraparesis
MeSH Terms: conditions — Quadriplegia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Assessment of upper limb variables (Experimental): Assessment of clinical variables of tetraplegics reach-and-grasp pattern
  Interventions: Other: Assessment of upper limb variables
- Training protocol (Experimental): Training with electrical stimulation of upper limb
  Interventions: Other: Training protocol

INTERVENTIONS:
Other: Assessment of upper limb variables — International Standards for Neurological and Functional Classification of Spinal Cord Injuries of American Spinal Injury Association (ASIA); Functional Independence Measure (FIM); The following kinematic variables of arm were studied: shoulder, elbow and wrist angles; percentage of time to peak velocity; movement time; peak velocity and movement smoothness (number of velocity peaks and index of curvature); Capabilities of Upper Extremity instrument (CUE); Spinal cord independence measure (SCIM II); electromyography (Clavicular portion of pectoralis major, long head of biceps brachii, anterior and posterior deltoid, triceps and wrist extensors).
  Arms: Assessment of upper limb variables
Other: Training protocol — The strengthening sessions consisted of 20 minutes of electrical stimulation on triceps, extensor carpi radialis longus, extensor digitorum communis, lumbricalis, flexor digitorum superficialis and opponens pollicis muscles. The functional training sessions was performed through movements the reach and palmar grasp with NMES of the several cylindrical and conical objects of different weights (30 minutes sessions).
  Arms: Training protocol

SUMMARY:
The aim of the study was to evaluate the tetraplegics movement strategies, assisted by Neuromuscular Electrical Stimulation (NMES), on the reach and palmar (RP) grasp to different weights objects.Tetraplegics had their RP grasp movement captured by four infrared cameras and 6-reflexive markers attached on the trunk and right arm, assisted or not by NMES, in the triceps, extensor carpi radialis longus, extensor digitorum communis, flexor digitorum superficialis, opponens pollicis and lumbricalis muscles. The grasp was made in three cylindrical objects (different diameters and weights) placed in trunk midline in an equivalent distance of the arm's length. The patients were able to reach and made palmar grasp in all cylinders using the stimulation sequences assisted by NMES.

DETAILED DESCRIPTION:
Prior to the kinematic captures, all patients selected in the study received 20 sessions of NMES therapy, twice a week, with 10 weeks of duration. The strengthening sessions plus training prior to the kinematic study of movement strategies has the objective to condition the paretic muscles to the functional activity.

Twenty sessions was divided in 10 sessions of strengthening and 10 sessions of the functional training of reaching and grasping assisted with electrical stimulation.

The strengthening sessions consisted of 20 minutes of electrical stimulation on triceps, extensor carpi radialis longus, extensor digitorum communis, lumbricalis, flexor digitorum superficialis and opponens pollicis muscles.

The functional training sessions was performed through movements the reach and palmar grasp with NMES of the several cylindrical and conical objects of different weights (30 minutes sessions). The NMES was used to facilitate movements of reach (triceps muscle), opening (extensor carpi radialis longus and extensor digitorum communis muscle), positioning (extensor carpi radialis longus, flexor digitorum superficialis and lumbricalis muscle), palmar grasp (extensor carpi radialis longus, flexor digitorum superficialis, opponens pollicis muscle) and releasing (extensor carpi radialis longus and extensor digitorum communis muscle). Since the temporal organization varied among tetraplegics, some of them required more time to some stages of the sequence.

For NMES, the eight-channel stimulator, controlled by a microcomputer was used with pulse frequency, 25 Hz; pulse duration, 300 milliseconds; on/off duration 2/2sec; maximum pulse width fixed at 250 microampere, and the amplitude individually adjusted to achieve the excitability threshold for each muscle. The amplitude was adjusted throughout the training, in order to produce the desired muscle contraction. This parameters was used in all of therapies and in the kinematic assessment. The stimulation was applied with self-adhesive surface electrodes taped to the skin.

For kinematic captures, the participants performed reach and grasp with the dominant arm (right), assisted and not assisted by NMES. The subjects had no restriction for trunk anterior shifting but for safety reasons were kept seating upright in their own daily use wheelchair (the one they were more adapted to) and the non-dominant arm (left) was left resting over the abdomen in an attempt to minimize the influence of the non evaluated member on postural control.

For the initial position, the dominant arm was held at the side of the trunk, with the elbow flexed at 90º and the forearm in neutral position on the table. Tetraplegic subjects were seated in front of a task-table with the cylinder on it. They were instructed to reach and grasp three different cylinders (object A :200g weight, 115 mm height, 40 mm diameter; object B: 270g, 115 mm e 50 mm; and object C: 480g, 115 mm e 60 mm), one at a time and bring it to the initial hand position.

The analysis of kinematic data was performed from the beginning of the movement (starting position), until the early return of hand position (with or without the cylinder). The cylinder was positioned in front of the subject sternum, with a distance equal to the arm's length (from the medial border of axilla to the distal wrist crease).

The subjects were asked to perform five repetitions of each task for all three cylinders, in a total of 15 repetitions assisted and 15 not assisted by NMES. Once the experiment started, the subject could not touch the table with the forearm, until the task was finished. The command used to start the experiment was "GO", and they were instructed to perform the movement naturally and not to worry about the velocity and time of duration. Patients were evaluated in the two situations (with and without NMES) with stimulation electrodes placed in the skin surface and the cables connected to the stimulator.

ELIGIBILITY:
Inclusion Criteria:

* tetraplegics (C4 to C7), complete or incomplete, traumatic lesion.

Exclusion Criteria:

* Neurological condition prior to spinal injury, orthopedic conditions in upper limb.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-12; Primary Completion 2006-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Upper limb Kinematics | change from baseline at twenty sessions - 5 weeks
  shoulder, elbow and wrist angles; percentage of time to peak velocity; movement time; peak velocity and movement smoothness (number of velocity peaks and index of curvature).

SECONDARY OUTCOMES:
ASIA | change from baseline at twenty sessions - 5 weeks
  Classification of injury by American Spinal Injury Association
SCIM II | change from baseline at twenty sessions - 5 weeks
  Spinal cord Independence measure
CUE | change from baseline at twenty sessions - 5 weeks
  capabilities of upper extremity
FIM | change from baseline at twenty sessions - 5 weeks
  Functional independence measure
Electromyography | change from baseline at twenty sessions - 5 weeks
  Clavicular portion of pectoralis major, long head of biceps brachii, anterior and posterior deltoid, triceps and wrist extensors

OTHER OUTCOMES:
demographic dates | baseline
  name, address, time since lesion, other injuries.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Cliquet Jr, PhD, Principal Investigator — University of Campinas

IPD SHARING:
Plan to Share IPD: No